CLINICAL TRIAL: NCT01099306
Title: Pharmacist - Physician Collaborative Approach to the Management of Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Eman Hammad, faculty of pharmacy / University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: JUaym8071383
Record Dates: First submitted 2010-04-05; First posted 2010-04-06 (Estimated); Last update posted 2010-04-06 (Estimated); Status verified 2009-03

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Pharmaceutical Services

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention (Active Comparator): pharmacist-physician collaborative approach to manage Metabolic syndrome
  Interventions: Other: Pharmaceutical care services
- control (No Intervention): physician only team to manage Metabolic syndrome

INTERVENTIONS:
Other: Pharmaceutical care services — Patients' metabolic components were assessed and managed collaboratively by focused care plan designed by the clinical pharmacist and approved by the physician.Pharmacist emphasized the change in lifestyle, particularly weight loss and physical activity as a first line therapy for at least 3 months, patients were started on drug therapy when needed as recommended by clinical guidelines.
  Arms: intervention

SUMMARY:
This study devised an experimental focused pharmaceutical care program, allowed a clinical pharmacist to work in a physician office to assess and manage patients' metabolic syndrome status and its individual components. This study described the clinical benefits of physician- clinical pharmacist interaction in achieving improved glycemic control, lipid and blood pressure measurements, involving medication, diet, physical activity and patient heath care counseling.

DETAILED DESCRIPTION:
A single blinded prospective randomized controlled trial conducted in family medicine outpatients clinics in Jordan. The study enrolled 199 patients met the National Cholesterol Education Program Adult Treatment Panel III (NCEP/ATPIII) criteria for the diagnosis of MS upon the time of enrollment. Patients were randomized into: 110 participants into the intervention arm (pharmacist-physician collaborative approach) and 89 into the control arm (physician only team). Only patients in the intervention arm were provided pharmacist recommendations and pharmaceutical care counseling.

ELIGIBILITY:
Inclusion Criteria:

* Meeting at least 3 of the 5 criteria for the National Cholesterol Education Program Adult Treatment Panel III (NCEP/ATPIII) for the diagnosis of Metabolic syndrome upon the time of enrollment. :

  1. Abdominal circumference >102 cm in males or >88 cm in females.
  2. HDL cholesterol < 40 mg/dl for males or < 50 mg/dl for females.
  3. Triglycerides ≥ 150 mg/dl.
  4. Blood pressure ≥ 130/85 mmHg or receiving hypertension treatment.
  5. Baseline glycemia ≥ 110 mg/dl.

Exclusion Criteria:

1. Patients with hypertensive urgency or emergency with BP more than (180/110).
2. Patients with recent stroke or myocardial infraction (within past 6 months).
3. Patients with Class III or IV Chronic heart Failure (CHF).
4. Patients with Unstable angina.
5. Patients with Serious renal or hepatic disease.
6. Pregnant patients.
7. Patients with Dementia or cognitive impairment.
8. If the patient is unable to provide informed written consent.

Ages: 32 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Improvements in metabolic syndrome status over the course of this study and absolute mean improvements in individual MS components. | 6 monthS
  Primary outcomes were specified as:
  * Fasting blood glucose < 110 mg/dl.
  * Body weight BMI < 25 kg/m2.
  * Waist circumference ≤ 102 cm (40 in) in men and ≤ 88 cm (35 inches) in women.
  * Serum triglycerides < 150 mg/dl.
  * HDL cholesterol ≥40mg/dl in men and ≥50mg/dl in women.
  * Blood pressure < 130/85 mm Hg or < 130/80 mm Hg when patients were diabetic.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Hammad, MSc, Principal Investigator — University of Jordan/ Faculty of Pharmacy; Abla Al bsoul, PhD, Study Director — University of Jordan/ Faculty of Pharmacy
Locations (1):
- family medicine clinic JUH, Amman, Amman Governorate, Jordan